CLINICAL TRIAL: NCT04882150
Title: A Phase 1, Randomized, Double-Blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BMS-986196 in Healthy Participants Including an Open-label Assessment of Food and Formulation Effects on the Relative Bioavailability of BMS-986196
Brief Title: A Study to Determine the Safety, Drug Levels and Drug Effects of BMS-986196 and Food and Formulation Effects on Relative Absorption Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM038-008
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy Participants
Keywords: Healthy participants; BMS-986196

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: SAD (Experimental): SAD = single ascending dose. Each participant will receive a single dose of BMS-986196 or placebo.
  Interventions: Drug: BMS-986196; Other: Placebo
- Part B: MAD (Experimental): MAD = multiple ascending dose. Each participant will receive multiple doses of BMS-986196 or placebo.
  Interventions: Drug: BMS-986196; Other: Placebo
- Part C: FE/Formul. (Experimental): FE/Formul. = food and formulation effects and relative absorption. Participants will receive two formulations of BMS-986196 (solution and suspension), each formulation with and without food.
  Interventions: Drug: BMS-986196

INTERVENTIONS:
Drug: BMS-986196 — Specified dose on specified days
Other: Placebo — Specified dose on specified days
  Arms: Part A: SAD; Part B: MAD

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, drug levels and drug effects of BMS-986196 in healthy participants. In addition, an evaluation of food and formulation effects on BMS-986196 absorption will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Women not of childbearing potential and men, ages 18 or local age of majority to 55 years, inclusive
* Healthy male and female non-Japanese participants without clinically significant deviation from normal in medical history, physical examination, electrocardiogram (ECG), and clinical laboratory determinations
* Body mass index (BMI) of 18 to 32 kg/m2, inclusive, and total body weight ≥ 50 kg

Exclusion Criteria:

* Known or suspected autoimmune disorder, including but not limited to rheumatoid arthritis, fibromyalgia, systemic lupus erythematosus, polymyalgia rheumatica, giant cell arteritis, Behcet's disease, dermatomyositis, MS, moderate to severe asthma, any autoimmune vasculitis, autoimmune hepatitis, or any other active autoimmune disease for which a participant requires medical follow-up or medical treatment
* Any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status
* Presence of any factors that would predispose the participant to develop infection
* A history of bacterial or fungal meningitis within 1 year prior to screening
* A history of intracranial or intraspinal bleeding
* Known intracranial space-occupying mass, including meningioma

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 24 days
Severity of AEs | Up to 24 days
Causality of AEs | Up to 24 days
Incidence of Serious Adverse Events (SAEs) | Up to 59 days
Severity of SAEs | Up to 59 days
Causality of SAEs | Up to 59 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 24 days
Incidence of clinically significant changes in vital signs: Respiratory rate | Up to 24 days
Incidence of clinically significant changes in vital signs: Blood pressure | Up to 24 days
Incidence of clinically significant changes in vital signs: Heart rate | Up to 24 days
Incidence of clinically significant changes in weight | Up to 24 days
Incidence of clinically significant changes in physical examination | Up to 24 days
Incidence of clinically significant changes in ECG parameters: QT interval | Up to 24 days
Incidence of clinically significant changes in ECG parameters: HR | Up to 24 days
Incidence of clinically significant changes in clinical laboratory values: Hematology tests | Up to 24 days
Incidence of clinically significant changes in clinical laboratory values: Clinical chemistry tests | Up to 24 days
Incidence of clinically significant changes in clinical laboratory values: Coagulation tests | Up to 24 days
Incidence of clinically significant changes in clinical laboratory values: Urinalysis tests | Up to 24 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0002, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome